CLINICAL TRIAL: NCT04562311
Title: The Efficacy and Safety of Chidamide Combined With Immunotherapy in Patients With Locally Advanced or Metastatic Urothelial Carcinoma Who Had Previously Received Platinum-based Chemotherapy:An Open, One-arm, Phase II Study
Brief Title: Chidamide With Immunotherapy for Patients With Locally Advanced or Metastatic Urothelial Carcinoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Head of UrologyDepartment,Sun Yat-sen University Cancer center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2020-192-01
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Bladder Cancer Stage IV
Keywords: Chidamide、Immunotherapy、Bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide with Immunotherapy (Experimental): Chidamide: 30mg orally BIW. Immunotherapy: tislelizumab,the fixed dose of 200 mg IV. Treatment cycles are repeated every 3 weeks.
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — Chidamide: 30mg orally BIW. Immunotherapy: tislelizumab,the fixed dose of 200 mg IV. Treatment cycles are repeated every 3 weeks.
  Other Names: Single-arm

SUMMARY:
Study of Chidamide Combined With Immunotherapy in Patients With Locally Advanced or Metastatic Urothelial Carcinoma Who Had Previously Received Platinum-based Chemotherapy

DETAILED DESCRIPTION:
Chidamide has been approved for the treatment of relapsed or refractory peripheral T-cell lymphoma in China (Chidamide,a novel histone deacetylase inhibitor). Tirelizumab,has been approved for the failure treatment of platinum-containing chemotherapy with high PD-L1 expression included locally advanced or metastatic Urothelial carcinoma in China(Tirelizumab,BGB-A317 is an investigational humanized IgG4 anti-PD-1 monoclonal antibody ).The aim of this study was to observe the efficacy and safety of Chidamide with Immunotherapy in patients with progression of platinum-based chemotherapy recurrent and metastatic Urothelial carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Age ≥18 years, < 75 years
* 2.Histopathological diagnosis of transitional cell carcinoma or urothelial carcinoma; It may be associated with other cell types such as small cell carcinoma, neuroendocrine carcinoma or squamous cell carcinoma, but the component should be mainly urothelial carcinoma
* 3.Patients with advanced urothelial carcinoma (inoperable or metastatic to lymph nodes or distant metastases) recurred or progressed during adjuvant therapy or advanced first-line platinum-based chemotherapy; Patients receiving secondary chemotherapy may be included, but more than 12 months from the end of the first chemotherapy to the beginning of the second chemotherapy; Subjects who receive neoadjuvant chemotherapy or adjuvant chemotherapy and who develop disease progression within 12 months of the last dose are considered to be receiving systemic chemotherapy in the context of cancer metastasis (disease progression is defined as any progression requiring a change in treatment regimen prior to treatment)
* 4.Measurable target lesion (without radiotherapy) : defined as having at least one lesion that can be accurately measured in at least one dimension (the longest diameter recorded), such as ≥15mm conventional technique or ≥10mm helical CT scan; Patients with bone metastases may also participate in the study, provided they also have a measurable non-osseous disease
* 5.Life expectancy is more than 3 months
* 6.ECOG performance status 0~2 (Karnofsky >= 60%)
* 7.Bone marrow, liver and renal function adequate: Blood routine examination: neutrophil count ≥2.0×109/L, PLT count ≥75×109/L, WBC count ≥3.0×109/L, hemoglobin concentration ≥90.0g/dL; Liver function: AST and ALT≤1.5 times the upper limit of normal value (ULN), alkaline phosphatase ≤1.5×ULN, TBIL≤ULN; Cr 1.5 x ULN or less
* 8.Left ejection fraction (LVEF) ≥50%, electrocardiogram (ECG) was generally normal, QTc interphase <0.44 seconds, and there were no signs or symptoms of heart failure
* 9. Acute toxicity caused by previous treatment is alleviated to level ≤1 (except hair loss)
* 10.The eligibility of patients receiving any drug or substance known or likely to affect cedaramide activity or pharmacokinetics will be determined after review by the principal investigator for a period of more than 6 weeks
* 11.Understand and be willing to sign written informed consent documents

Exclusion Criteria:

* 1.Patients who received chemotherapy (nitrosourea or mitomycin C for 6 weeks) within 4 weeks before the study began, or who did not recover from adverse events due to drug use more than 4 weeks in advance
* 2.Patients shall not receive any other anticancer drugs or clinical trial drugs during the clinical trial period (local palliative radiotherapy other than the target lesion may be accepted)
* 3.Patients with brain metastases
* 4.A history of allergic reactions to compounds that are chemically or biologically similar to cedarbenamine; These compounds include sodium butyrate, Trichostatin A (TSA), Trapoxin (TPX), MS-27-275, and Depsipeptide
* 5.Treatment of Urothelial carcinoma with more than two lines or above cytotoxic chemotherapy regiments
* 6.Uncontrolled underlying concomitant diseases, including but not limited to persistent or active infections, symptomatic congestive heart failure, unstable angina, arrhythmia, or psychiatric/social conditions, may limit compliance with study requirements
* 7.Pregnant women are excluded and should stop breastfeeding if they receive treatment during lactation in the study
* 8.Long-term use of immunosuppressive agents after organ transplantation; Patients with autoimmune diseases; Patients who are taking immunosuppressive drugs
* 9.HIV positive or have other immunodeficiency diseases
* 10.Combined with other active malignancies (i.e., changes in treatment required within the past 24 months). Only patients with skin cancer that has been treated within the past 24 months and has been completely cured are allowed to be enrolled. Localized prostate cancer with Gleason score of 6 (treated or untreated but monitored within the past 24 months); Localized prostate cancer with a Gleason score of 3+4 that was treated more than 12 months prior to full study screening and was completely cured
* 11.Live virus vaccine is administered within 30 days of initial administration
* 12.Patients should not take valproic acid for at least 2 weeks before entering the study
* 13.Due to psychological, social, family, geographical and other reasons can not cooperate with regular follow-up observers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate（ORR） | up to 2 years
  Objective Response Rate（ORR）by RECIST 1.1,the total proportion of patients with complete response（CR）, partial response（PR）

SECONDARY OUTCOMES:
Disease Control Rate （DCR） | up to 2 years
  the total proportion of patients with complete response（CR）, partial response（PR）and Stable Disease（SD）
Progression-free survival(PFS) | up to 2 years
  Time from treatment until disease progression or death
Overall survival(OS) | up to 2 years
  Time from treatment until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jianfang Zhou, Study Chair — Sun Yat-sen University
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shi Y, Jia B, Xu W, Li W, Liu T, Liu P, Zhao W, Zhang H, Sun X, Yang H, Zhang X, Jin J, Jin Z, Li Z, Qiu L, Dong M, Huang X, Luo Y, Wang X, Wang X, Wu J, Xu J, Yi P, Zhou J, He H, Liu L, Shen J, Tang X, Wang J, Yang J, Zeng Q, Zhang Z, Cai Z, Chen X, Ding K, Hou M, Huang H, Li X, Liang R, Liu Q, Song Y, Su H, Gao Y, Liu L, Luo J, Su L, Sun Z, Tan H, Wang H, Wang J, Wang S, Zhang H, Zhang X, Zhou D, Bai O, Wu G, Zhang L, Zhang Y. Chidamide in relapsed or refractory peripheral T cell lymphoma: a multicenter real-world study in China. J Hematol Oncol. 2017 Mar 15;10(1):69. doi: 10.1186/s13045-017-0439-6. PMID 28298231
- [Background] Li Y, Chen K, Zhou Y, Xiao Y, Deng M, Jiang Z, Ye W, Wang X, Wei X, Li J, Liang J, Zheng Z, Yao Y, Wang W, Li P, Xu B. A New Strategy to Target Acute Myeloid Leukemia Stem and Progenitor Cells Using Chidamide, a Histone Deacetylase Inhibitor. Curr Cancer Drug Targets. 2015;15(6):493-503. doi: 10.2174/156800961506150805153230. PMID 26282548
- [Background] Zhang L, Han Y, Jiang Q, Wang C, Chen X, Li X, Xu F, Jiang Y, Wang Q, Xu W. Trend of histone deacetylase inhibitors in cancer therapy: isoform selectivity or multitargeted strategy. Med Res Rev. 2015 Jan;35(1):63-84. doi: 10.1002/med.21320. Epub 2014 Apr 29. PMID 24782318
- [Background] Bellmunt J, de Wit R, Vaughn DJ, Fradet Y, Lee JL, Fong L, Vogelzang NJ, Climent MA, Petrylak DP, Choueiri TK, Necchi A, Gerritsen W, Gurney H, Quinn DI, Culine S, Sternberg CN, Mai Y, Poehlein CH, Perini RF, Bajorin DF; KEYNOTE-045 Investigators. Pembrolizumab as Second-Line Therapy for Advanced Urothelial Carcinoma. N Engl J Med. 2017 Mar 16;376(11):1015-1026. doi: 10.1056/NEJMoa1613683. Epub 2017 Feb 17. PMID 28212060